CLINICAL TRIAL: NCT02286167
Title: The Feasibility and Biologic Effect of a Modified Atkins-based Intermittent Fasting Diet in Patients With Glioblastoma (GBM)
Brief Title: Glioma Modified Atkins-based Diet in Patients With Glioblastoma
Acronym: GLAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00037347
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2019-08

CONDITIONS: Glioblastoma Multiforme
Keywords: modified-Atkins diet; ketogenic diet; central nervous system malignancy; glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm diet (Other): Intermittent, modified Atkins diet
  Interventions: Other: Diet modification

INTERVENTIONS:
Other: Diet modification — All patients will be participate in the intermittent, modified Atkins diet

SUMMARY:
The primary goal of this study is to assess the feasibility and biologic activity of a modified Atkins-based diet combined with short-term intermittent fasting, a GLioma Atkins-based Diet (GLAD), in patients with central nervous system GBM.

DETAILED DESCRIPTION:
Malignant gliomas have a high glycolytic rate and are dependent on glucose for energy metabolism. This so called "Warburg effect" or the reliance of central nervous system (CNS) tumor cells on glucose utilization through glycolysis has been identified as a potential therapeutic target in cancer metabolism. Preclinically, reduced cerebral glucose via calorie restriction has been repeatedly associated with tumor reduction and improved survival in glioma animal models. Such work has led to several early clinical studies evaluating the ketogenic diet (KD) in patients with recurrent GBM.

The modified Atkins diet (MAD) is designed to provide a more palatable, less restrictive but effective alternative to the strict KD, particularly for adults. The MAD does not require inpatient admission for initial fast, weight of foods, or severe dietary restrictions and is generally well tolerated, easier to administer, and more practical for adults. The MAD lacks calorie restriction, an important component to dietary therapies in preclinical investigations. Emerging evidence also suggests that short term fasting may provide superior anti-cancer activity to long term calorie restriction and that these benefits have been observed without substantial weight loss that can be observed with longer term calorie restriction.

In glioma patients, a diet therapy that combines the broad clinical application of the MAD with the caloric impact of short-term intermittent fasting is therefore optimal. Moreover, initiation of this diet when the cancer has already undergone induction therapy and is clinically and radiographically stable, may provide the optimal time for metabolic intervention to prevent recurrence or progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a clinical and histopathologic diagnosis of GBM, have completed >80% of prescribed concurrent radiation therapy and adjuvant temozolomide without CTCEA grade 3 or 4 toxicity, and be greater than 7 months from the time of completion of concurrent chemoradiotherapy.
2. Karnofsky performance status >/= 60.
3. Patients must be at least 18 years of age.
4. Patients must be eligible to undergo a ketogenic or Atkins based diet according to baseline body mass index (BMI, see exclusion criteria), comorbid medical conditions (see exclusion criteria), and baseline laboratory assessment (see exclusion criteria).
5. Patients must be of appropriate mental capacities with sufficient social support so as to be able to complete required study activities (i.e. diet record, etc) and able to provide written informed consent.

Exclusion Criteria:

1. Patients with a history of a metabolic disorder including documented defect in urea metabolism (including documented history of gout), carnitine deficiency (primary carnitine deficiency, carnitine palmitoyltransferase I or II deficiency, carnitine translocase deficiency), fatty acid metabolism, beta-oxidation defects, pyruvate carboxylase deficiency, mitochondrial function, porphyria, or nephrolithiasis.
2. Severe acute infection.
3. BMI > 35.0 or BMI < 20.0.
4. Active bowel obstruction, ileus, or active or remote pancreatitis.
5. Clinically significant heart failure (NYHA >2), recent myocardial infarction, or symptomatic atrial fibrillation.
6. Clinically significant renal disease (creatinine >2.0 mg/dL, urea >100 mg/dL).
7. Clinically significant hepatic dysfunction (alanine or aspartate aminotransferase >7 times the upper limit of normal).
8. Patients with insulin-dependent diabetes mellitus.
9. Conditions that may increase the risk of the diet or significantly reduce compliance (i.e. cognitive impairment, frank dementia, etc).
10. Other concurrent experimental therapies.
11. Milk allergy.
12. Treatment with the modified Atkins diet (MAD) for any cause within the 9 months prior to study enrollment
13. Patient inability to complete baseline screening 3-day diet record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of intermittent modified Atkins diet in patients with GBM assessed by percent of patients able to remain on the diet and achieve nutritional goals | 8 weeks per patient
  Percent of patients able to remain on the diet and achieve nutritional goals as defined by cumulative assessment of diet records collected at weeks 4, 6, and 8 with a 60% completion defined as a positive results

SECONDARY OUTCOMES:
Biologic activity measured by pre- and post-study cerebral glutamate and glutamine concentrations assessed by MRS. | 8 weeks per patient
  Measured by pre- and post-study cerebral glutamate and glutamine concentrations assessed by MRS.
Tolerability assessed by percent of patients who have an adverse reaction of any grade attributed to the diet of possible, probable, or definite | 8 weeks per patient
  Percent of patients who have an adverse reaction of any grade attributed to the diet of possible, probable, or definite
Dietary Activity | 8 weeks per patient
  Dietary compliance will be assessed by serial changes in serum glucose, ketones, weight trajectory, body fat composition, change in seizure frequency without AED adjustment

CONTACTS AND LOCATIONS:
Overall Officials: Roy E. Strowd, MD, Principal Investigator — Wake Forest University Health Sciences; Jaishri O. Blakeley, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Wake Forest School of Medicine, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Schreck KC, Hsu FC, Berrington A, Henry-Barron B, Vizthum D, Blair L, Kossoff EH, Easter L, Whitlow CT, Barker PB, Cervenka MC, Blakeley JO, Strowd RE. Feasibility and Biological Activity of a Ketogenic/Intermittent-Fasting Diet in Patients With Glioma. Neurology. 2021 Aug 31;97(9):e953-e963. doi: 10.1212/WNL.0000000000012386. Epub 2021 Jul 7. PMID 34233941

DOCUMENTS (1):
  • Informed Consent Form (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT02286167/ICF_000.pdf